CLINICAL TRIAL: NCT05428020
Title: The Use of a Routine Indwelling Urinary Catheter in Patients Receiving Neuraxial Anesthesia for Elective Total Joint Arthroplasty
Brief Title: RCT Foley Catheter Study for Elective TJA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Responsible Party: Principal Investigator, Craig J Della Valle, MD, Professor of Orthopedic Surgery, Chief Division of Adult Reconstruction, Rush University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 19123101
Record Dates: First submitted 2022-06-16; First posted 2022-06-22 (Actual); Results first posted 2023-08-03 (Actual); Last update posted 2023-08-03 (Actual); Status verified 2023-07

CONDITIONS: Postoperative Urinary Retention; Total Hip Arthroplasty; Total Knee Arthroplasty
Keywords: total knee arthroplasty; total hip arthroplasty; indwelling catheter; Foley catheter; arthroplasty
MeSH Terms: interventions — Urinary Catheterization

STUDY DESIGN:
Who Masked: Participant
Masking Description: The participant (patient) will be blinded to whether they are receiving a short-term foley catheter or no foley.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Indwelling foley catheter (Experimental): Short-term indwelling foley catheter
  Interventions: Device: Indwelling foley catheter
- No Foley catheter (Placebo Comparator): No foley catheter
  Interventions: Other: No foley catheter

INTERVENTIONS:
Device: Indwelling foley catheter — short-term indwelling catheter inserted in the operating room prior to surgery, removed upon arrival to the floor from post-anesthesia care unit (approx 2-3 hours after surgery).
  Other Names: foley
  Arms: Indwelling foley catheter
Other: No foley catheter — No foley catheter is placed for surgery
  Arms: No Foley catheter

SUMMARY:
Urinary retention is a known complication following surgical procedures, with a theoretical increased risk in patients receiving neuraxial anesthesia due to a decreased ability to sense bladder distension. Urinary retention is associated with adverse events including bladder atony, increased post void residuals, and postoperative urinary tract infection. Treatment of urinary retention involves intermittent or indwelling urinary catheter placement, both of which are associated with an increased prevalence of postoperative urinary tract infection.

There currently is no consensus whether the use of a urinary catheter in elective joint arthroplasty with neuraxial anesthesia decreases the risk of urinary retention. The prevalence of retention reported in the literature varies widely with reports anywhere from 0% to 75% in patients with early removal of a catheter or after procedures performed without a catheter.

The goal of this study is to determine whether the routine use of an indwelling urinary catheter decreases the rate of postoperative urinary retention in patients undergoing elective joint arthroplasty.

DETAILED DESCRIPTION:
Study Design

Treatment Groups:

Group 1 (Control): Short term urinary catheter- Patient will receive a urinary catheter at the time of the surgery. The urinary catheter will be removed upon arrival to the orthopedic floor post operatively. Patients will subsequently be monitored for urinary retention according to the Rush University Medical Center urinary retention protocol.

Group 2 (Experimental): No urinary catheter- Patients will not receive a urinary catheter at time of surgery. They will be monitored for urinary retention according to the Rush University Medical Center urinary retention protocol

Sample Size Calculation Based on a randomized controlled trial published by Miller et al in 2013, to detect a clinically significant difference of 7%, we would need 194 patients per group, or 388 patients. Assuming a drop-out rate of 10%, a total of 432 patients will be required. An interim analysis will be performed once half of this total is enrolled.

Urinary retention protocol:

Patients will be monitored closely for urinary retention according to current Rush University Medical Center Urinary Retention Protocol. After removal of catheter (control group) or from arrival in post-anesthesia care unit (experimental group), patients will be given 4 hours to void a volume corresponding to 30ml/hour. If the patient fails to do so, they will be bladder scanned. Bladder scan results of 450ml or greater will result in one time straight catheterization. If bladder scan shows 150 ml to 349 ml of urine, patients will be given an additional 4 hours to void and a repeat bladder scan will be performed. If unable to void at this point and/or bladder volume is >450, patient will receive a one time straight catheterization.

If bladder scan shows 350 ml to 449 ml of urine, patients will be given an additional 2 hours to void and a repeat bladder scan performed. If unable to void at this point and/or bladder volume is >450, patient will receive a one time straight catheterization.

If patients require a straight catheterization, they will be monitored with bladder scan according to protocol and a second straight catheterization will be performed if necessary. At time of second straight catheterization, a urinalysis will be sent. If patient requires a third straight catheterization, a urology consult will be placed according to protocol and patient will either receive an indwelling urinary catheter or intermittent straight catheterization with urology follow up.

Demographics, Patient Specifics Age, sex, short form 12 scores, american society of anesthesia (ASA) score, medical co-morbidities, weight, height, length of hospitalization, BMI, history of benign prostatic hypertrophy, presence of preoperative urinary tract infection (diagnosed during preadmission testing), intravenous fluids given during surgery, operating room time, estimated blood loss, length of hospital stay, discharge destination (home versus rehabilitation facility), time to mobilization postoperatively, and length of urinary catheter usage.

At the time of enrollment in the study, patients will be given a urinary history questionnaire known as the International Prostate Symptom Score (I-PSS) and be asked about history of urinary retention, history of incontinence, and history of polyuria to screen for preexisting urinary issues. Patients will receive a urinalysis as part of preoperative testing to screen for presence of urinary tract infection. Patients will receive standardized multimodal analgesic regimen that is utilized at Rush University Medical Center for patients undergoing a total joint replacement for perioperative and postoperative pain management. Modifications will be made on a case by case basis as is currently the standard practice (for example, allergy, intolerance, or medical contraindication such as acute kidney injury to NSAID use)

ELIGIBILITY:
Inclusion Criteria:

* Any patient >18 years of age scheduled for an inpatient primary hip or knee replacement

Exclusion Criteria:

* Patients with a known history of prostate, urological or kidney surgery
* Patients where close monitoring of urine output are necessary during the perioperative period (renal disease, renal failure, chronic indwelling urinary catheter)
* Patients with a history of urinary incontinence
* Patients undergoing a revision total knee or total hip arthroplasty
* Patients requiring indwelling continuous epidural anesthesia
* Patients with a preexisting urinary tract infection, as diagnosed on preoperative screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 388 (Actual)
Dates: Start 2020-11-16 (Actual); Primary Completion 2022-05-25 (Actual); Study Completion 2022-11-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Craig Della Valle, MD, Principal Investigator — Rush University Medical Center
Locations (1):
- Rush University medical Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No
Abstract and Manuscript write up upon completion of study

REFERENCES:
- [Background] Balderi T, Carli F. Urinary retention after total hip and knee arthroplasty. Minerva Anestesiol. 2010 Feb;76(2):120-30. PMID 20150853
- [Background] Lo E, Nicolle L, Classen D, Arias KM, Podgorny K, Anderson DJ, Burstin H, Calfee DP, Coffin SE, Dubberke ER, Fraser V, Gerding DN, Griffin FA, Gross P, Kaye KS, Klompas M, Marschall J, Mermel LA, Pegues DA, Perl TM, Saint S, Salgado CD, Weinstein RA, Wise R, Yokoe DS. Strategies to prevent catheter-associated urinary tract infections in acute care hospitals. Infect Control Hosp Epidemiol. 2008 Oct;29 Suppl 1:S41-50. doi: 10.1086/591066. No abstract available. PMID 18840088
- [Background] Farag E, Dilger J, Brooks P, Tetzlaff JE. Epidural analgesia improves early rehabilitation after total knee replacement. J Clin Anesth. 2005 Jun;17(4):281-5. doi: 10.1016/j.jclinane.2004.08.008. PMID 15950853
- [Background] Borghi B, Agnoletti V, Ricci A, van Oven H, Montone N, Casati A. A prospective, randomized evaluation of the effects of epidural needle rotation on the distribution of epidural block. Anesth Analg. 2004 May;98(5):1473-8, table of contents. doi: 10.1213/01.ane.0000111113.45743.b8. PMID 15105234
- [Background] Miller AG, McKenzie J, Greenky M, Shaw E, Gandhi K, Hozack WJ, Parvizi J. Spinal anesthesia: should everyone receive a urinary catheter?: a randomized, prospective study of patients undergoing total hip arthroplasty. J Bone Joint Surg Am. 2013 Aug 21;95(16):1498-503. doi: 10.2106/JBJS.K.01671. PMID 23965700
- [Background] Anger J, Lee U, Ackerman AL, Chou R, Chughtai B, Clemens JQ, Hickling D, Kapoor A, Kenton KS, Kaufman MR, Rondanina MA, Stapleton A, Stothers L, Chai TC. Recurrent Uncomplicated Urinary Tract Infections in Women: AUA/CUA/SUFU Guideline. J Urol. 2019 Aug;202(2):282-289. doi: 10.1097/JU.0000000000000296. Epub 2019 Jul 8. PMID 31042112
- [Background] Darbyshire D, Rowbotham D, Grayson S, Taylor J, Shackley D. Surveying patients about their experience with a urinary catheter. Int J of Uro Nursing 2016;10(1):14-20.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Indwelling Foley Catheter | No Foley Catheter
Started | 194 | 194
Completed | 194 | 194
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Indwelling Foley Catheter | No Foley Catheter | Total
Number analyzed (Participants) | 194 | 194 | 388
Age, Continuous [Mean (Full Range); unit: years] | 67.36 [30.53 to 88.81] | 67.12 [41.52 to 90.18] | 67.24 [30.53 to 90.18]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 125 | 120 | 245
  Male | 69 | 74 | 143
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White/caucasion | 144 | 158 | 302
  Race: Black/African American | 46 | 32 | 78
  Race: Asian | 4 | 4 | 8
Region of Enrollment [Number; unit: participants]
  United States | 194 | 194 | 388

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Who Developed Postoperative Urinary Retention (POUR), Unable to Void a Volume Greater Than or Equal to 30ml/hr
Description: All patients were monitored per hospital protocol for urinary retention. After removal of catheter (control group) and those without (experimental group) upon arrival in the PACU (post anesthesia care unit), patients were given 4 hours to void a volume corresponding to 30ml/hour. If the patient failed to do so, they would have their bladder scanned. Bladder scanned results were all reported by 4 hours after surgery. Patients inability to void a volume corresponding to 30ml/hour AND after straight catheterization (per hospital protocol), meant they developed POUR following surgery.
Time Frame: While inpatient following surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Indwelling Foley Catheter | No Foley Catheter
Number analyzed (Participants) | 194 | 194
Participants | 4 | 5

2. Secondary Outcome: Urinary Tract Infections (UTI) as Complication up to 3 Weeks Following Total Joint Arthroplasty
Description: Patients who are treated following Total Joint Arthroplasty for UTI
Time Frame: up to 3 weeks after surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Indwelling Foley Catheter | No Foley Catheter
Number analyzed (Participants) | 194 | 194
Participants | 3 | 1

3. Secondary Outcome: Straight Catheterization Required While Inpatient Following Total Joint Arthroplasty
Description: Patient requires 1 or more straight catheterization while inpatient, due to inability to void 30ml/hr during the patient's hospital stay. Straight catheterizations are performed by placing an indwelling catheter when indicated by retention of ≥450 mL on bladder scans. Bladder scans are performed per hospital protocol for patients unable to void a volume of 30ml/hr in the first 4 hours following surgery. If bladder shows 150 ml to 349 ml of urine, patients are given another 4 hours to void, followed by a repeat bladder scan. If unable to void at that time, or bladder volume is >450ml, patient will receive one-time catheterization.
  If bladder scan shows 350 ml to 449 ml of urine, they will be given 2 hours to void and repeat bladder scan. If unable to void or bladder volume is >450 ml, patient receives one time catheterization.
  If patient receives straight catheterization, they're monitored according to protocol and a second straight catheterization is done if necessary.
Time Frame: While inpatient at hospital, immediately following surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Indwelling Foley Catheter | No Foley Catheter
Number analyzed (Participants) | 194 | 194
Participants | 10 | 14

ADVERSE EVENTS:
Time Frame: 3 months following surgery, patients are followed for 90-day complications.
Arm/Group | Indwelling Foley Catheter | No Foley Catheter
All-Cause Mortality (participants affected / at risk) | 0/194 | 0/194
Serious Adverse Events (participants affected / at risk) | 0/194 | 0/194
Other Adverse Events (participants affected / at risk) | 0/194 | 0/194

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-10-07): https://cdn.clinicaltrials.gov/large-docs/20/NCT05428020/Prot_SAP_001.pdf